CLINICAL TRIAL: NCT06889766
Title: A Phase I Study Evaluating Safety and Feasibility of Redirected Autologous T Cells Expressing a High Affinity TCR Specific for NY-ESO-1 (LauT-1) in Patients With Advanced Melanoma and Sarcoma
Brief Title: NY-ESO-1-redirected T Cells in Patients With Advanced Melanoma and Sarcoma
Acronym: LauT1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Bernhard Gentner, Professor of Immuno-Oncology, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0026-NYESO1-2023
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Advanced Melanoma; Melanoma Metastatic; Sarcoma
Keywords: NY-ESO-1; LauT-1; TCR redirected T cell; metastatic melanoma; Sarcoma; autolog T-cell
MeSH Terms: conditions — Sarcoma; Melanoma | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: This study is a single center, Phase I, feasibility and safety trial without comparative arms, enrolling up to 9 patients in 2 dose cohorts.
  The safety run-in cohort will follow a 3+3 algorithm. The first 3 patients will be recruited sequentially and receive a target dose of 2x10^9 total cells (cohort 1), or a minimum of 3x10^8 NY-ESO-1 I53F transduced T cells (LauT-1).
  In the absence of treatment-limiting toxicity in the safety cohort, then up to 6 additional patients will receive the maximum number of LauT-1 product resulting from the manufacturing run, with an upper limit of 1x10^10 total cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study (Other)
  Interventions: Biological: NY-ESO-1 TCR redirected autologous T cell product; Radiation: Low-dose irradiation; Drug: Non-myeloablative lymphodepleting chemotherapy

INTERVENTIONS:
Biological: NY-ESO-1 TCR redirected autologous T cell product — Ex vivo expanded autologous CD4+/CD8+ cells expressing the transgenic TCR I53F recognizing NY-ESO-1 peptides presented on tumor cells in the context of HLA-A*02. The LauT-1-ACT infusion contains a minimum of 3x10^8 transduced cells (i.e. CD3+vβ13.1+) and a maximum of 1x10^10 total cells.
  Other Names: LauT-1
Radiation: Low-dose irradiation — 1Gy will be administered using tomotherapy (Accuray) to all irradiable lesions.
Drug: Non-myeloablative lymphodepleting chemotherapy — Fludarabine (30 mg/m2 x 4 days, from D-6 to D-3) and cyclophosphamide (2400 mg/ m2 x 2 days, on days -6 and -5) are administered as an IV infusion. The cyclophosphamide dose may be reduced to 1800mg/m2 on days -6 and -5, if the patient has previously been exposed to significant cumulative doses of chemotherapy)

SUMMARY:
A single center, Phase I clinical trial to demonstrate safety and efficacy of LauT-1, autologous "New York Esophageal Squamous Cell Carcinoma-1 T-Cell Receptor (NY-ESO-1 TCR)-directed T cells in combination with non-myeloablative (NMA) lymphodepleting chemotherapy and low dose irradiation (LDI) in patients with NY-ESO-1 positive sarcoma and melanoma.

DETAILED DESCRIPTION:
In this study, the investigators target the cancer testis antigen NY-ESO-1, which is highly expressed in a subset of sarcoma and melanoma but is largely absent in normal tissues. The affinity enhanced, Human Leukocyte Antigen - A2 (HLA-A2) restricted I53F T-cell receptor (TCR) used in this study is derived from a TCR originally isolated from a melanoma patient and recognizes the 157-165 epitope of the NY-ESO-1 protein with high affinity. The patients' own T-cells will be isolated, then genetically modified to express the I53F NY-ESO-1 TCR and expanded to generate the product "LauT-1", which is reinfused into the patients following lymphodepleting chemotherapy (LDCT) and low dose tumor irradiation (LDTI). LDCT allows maximal expansion of the infused T cells, and LDTI has been shown to inflame the tumor microenvironment in preliminary clinical data from recent studies, which may be useful to enhance T-cell infiltration and provide co-stimulatory signals within the tumor microenvironment, thereby maximising the chance to detect and potentially eliminate NY-ESO-1 expressing tumor cells.

In the current phase I study, the investigators assess the safety and feasibility of adoptive transfer of LauT-1 after LDCT and LDTI in HLA-A*0201 and/or HLA-A*0205 positive patients with advanced melanoma or sarcoma expressing NY-ESO-1. The experimental products are given initially to a group of 3 patients (safety cohort). If safe, the product may be given at a higher dose to 6 additional study participants (expansion cohort).

Procedures:

After confirming the expression of the NY-ESO-1 protein in at least 50% of the tumor cells and the presence of a permissive HLA allele during the pre-screeening procedure, patients eligible for the study will be undergo medical screening and registration to the study, followed by leukapheresis for the collection of autologous white blood cells (T lymphocytes) for the production of the gene-modified LauT-1 product. After successful leukapheresis, patients are allowed to receive a bridging therapy at the discretion of the PI/treating physician.

If all conditions are met and LauT-1 production is completed, the patient will start intravenous (IV) non-myeloablative lymphodepleting chemotherapy (LDCT) composed of fludarabine and cyclophosphamide. Both treatments will be started on the same day. Fludarabine will be given for four days, and cyclophosphamide for 2 days. LDTI will be administered as a single dose on Day 0 to all irradiable lesions using tomotherapy.

On D0, patients will receive NY-ESO-1 TCR T cell infusion, intravenously. Supportive care will be given as needed during the whole treatment period, and patients will be discharged according to institutional practice standards once they have achieved hematologic recovery, in the absence of other reasons for hospitalization. Patients will then be followed weekly in the outpatient clinic until the end of the Treatment-Limiting Toxicity (TLT) period, which extends from the first day of lymphodepleting chemotherapy to D30 after LauT-1 infusion. After the end of treatment visit, patients will be followed at the outpatient clinic by clinical & laboratory examination, as well as tumor assessment according to study schedule.

ELIGIBILITY:
Inclusion criteria at pre-screening step-1 1) Patients with histologically confirmed advanced or metastatic cutaneous melanoma or any type of sarcoma.

Inclusion criteria at pre-screening step-2

1) Immunohistochemically documented NY-ESO-1 expression, defined as ≥ 1+ expression on either archival or fresh tumor tissue by immunohistochemistry, in ≥50% of the sampled tumor tissue.

Inclusion criteria at screening

1. Patients with sarcoma, who have received at least one line of standard therapy (if available) and failed to respond, progressed or were intolerant to that therapy, will be eligible. If the participant refuses or is, in the opinion of the investigator, ineligible for these treatments, the reason must be documented in the medical record.
2. Patients with metastatic melanoma:

   1. Without proto-oncogene B-Raf (BRAF) mutation who have received at least one line of standard therapy and failed to respond, progressed or were intolerant to that therapy, will be eligible. If the participant refuses or is, in the opinion of the investigator, ineligible for these treatments, the reason must be documented in the medical record.
   2. With BRAF mutation who have received at least two lines of standard therapy and failed to respond, progressed or were intolerant to that therapy, will be eligible. If the participant refuses or is, in the opinion of the investigator, ineligible for these treatments, the reason must be documented in the medical record.
3. Patient must be HLA-A*0201 and/or HLA-A*0205 positive, as identified by high-resolution genomic deoxyribonucleic acid (DNA) typing of the HLA-A locus.
4. Age ≥ 18 years
5. Able to undergo apheresis
6. At least one lesion accessible to biopsy for translational research (TR) at D30, without putting the patient at unusual risk.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
8. Life expectancy of greater than 12 weeks.
9. Radiologically measurable disease (as per RECIST v1.1).
10. Adequate organ function

Exclusion Criteria:

1. Patients with an active second malignancy
2. Patients with symptomatic and/or untreated brain metastases, as well as leptomeningeal carcinomatosis. Patients with definitively treated brain metastases will be considered for enrolment after agreement with the Principal Investigator, as long as lesions are stable, there are no new brain lesions, and the patient does not require chronic corticosteroid treatment.
3. History of idiopathic pulmonary fibrosis or evidence of active pneumonitis (any origin). History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
4. History of recent myocardial infarction, or unstable angina, within six months prior to enrolment
5. Patients with prior allogeneic stem cell transplantation or organ transplantation
6. Active severe systemic infections within 2 weeks prior to apheresis
7. Patient requiring regular systemic immunosuppressive therapy. All immunosuppressive medications including but not limited to steroids, mycophenolate mofetil, azathioprine, methotrexate, thalidomide, and anti-Tumor Necrosis Factor-alpha (TNF-alpha) agents must have been discontinued at least 2 weeks before apheresis .
8. History of severe immediate hypersensitivity reaction to any of the agents/ excipients of the study products.
9. Women who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
10. Subjects, for whom there are concerns that they will not reliably comply with the requirements for contraception, should not be enrolled into the study.
11. Any serious underlying medical condition that could interfere with study medication and potential adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the incidence of treatment emergent adverse events | 90 days
  Safety of LauT-1 plus LDI after lymphodepleting chemotherapy will be established by classifying the observed toxicities by the MedDRA system and grading them using the National Cancer Institute (NCI) Common Toxicity Criteria (CTCAE Version 5.0) or American Society for Transplantation and Cellular Therapy (ASTCT) Cytokine Release Syndrom (CRS) consensus grading, as applicable.
Feasibility as measured by the rates of production failure and drop-outs before infusion | From start of LauT-1 production to treatment at 3 weeks
  Feasibility of LauT-1 production and administration will be evaluated as the number of cases for whom production of LauT-1 was successful (product was released based on specification criteria), and number of patients who receive LauT-1 at the intended dose according to the assigned dose-level, among all registered patients

SECONDARY OUTCOMES:
Long term safety as measured by the incidence of TEAE | 24 months
  Evaluated by documenting clinical and laboratory abnormalities, absence of replication-competent lentivirus, absence of abnormal clonal proliferation and organ toxicity using the MedDRA classification and the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0).
2. Objective response rate (ORR) | 90 days for each patient
  Evaluated according to Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1), overall and by cohort. ORR is defined as the rate of patients with best overall response objective response (Complete Response (CR) or Partial Response (PR)) within the first 90 days following LauT-1 infusion.
Disease control rate (DCR) | 2 years
  Evaluated according to RECIST 1.1, overall and by cohort. DCR is defined as the rate of patients with best overall response stable disease (for at least 3 months) or objective response (CR or PR) across all assessment time-points during the period from enrollment to termination of follow-up or progression (if it occurs before the end of follow-up).
Progression-free survival (PFS) | 24 months
  Is evaluated at 6, 12 and 24 months, where PFS is defined as the time from enrolment until objective tumor progression (using RECIST criteria) or death, if not documented progression.
Overall survival (OS) | 24 months
  OS rate is defined as the time from enrolment until death from any cause. If there is no death date, the patient will be censored at the last day the patient was known to be alive.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud